CLINICAL TRIAL: NCT04810975
Title: Strength Training Effects on Musculoskeletal Health, Melatonin, Rest-activity Rhythms and Quality of Life: Muscle:Time Study
Brief Title: Strength Training Effects on Musculoskeletal Health
Acronym: Muscle:Time
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duquesne University (Other)
Collaborators: Jaquish Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-12-15
Record Dates: First submitted 2021-03-18; First posted 2021-03-23 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Musculoskeletal Diseases
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The effect of exercise A on musculoskeletal health (Other)
  Interventions: Device: Muscle Strength Training
- The effect of exercise B on musculoskeletal health (Other)
  Interventions: Device: Muscle Strength Training

INTERVENTIONS:
Device: Muscle Strength Training — Strength training occurring specific exercise regimens using Exercise Equipment A or B

SUMMARY:
The objective here is to assess the efficacy of variable resistance muscle training on bone, sleep parameters and quality of life in healthy populations of men and women age 30 or older.

ELIGIBILITY:
Inclusion Criteria:

* 30 years or older (males or females)
* Baseline strength (e.g., can lift an office chair with no problems)
* Be willing to participate in a 6-month RCT
* Be willing to conduct daily muscle training exercises
* Be willing to maintain a food diary
* Be willing to consume ~2.2g/kg body weight daily
* Be willing to submit specimens and conduct tests 3 times over 6 months (0, 3 and 6 months)

Exclusion Criteria:

* those who consume vegan or vegetarian diets
* people with conditions like hypertension and uncontrolled non-medicated blood pressure; cardiovascular disease/heart failure (e.g., arrhythmias, unstable angina, congestive heart failure)
* COPD
* drugs that may increase fall risk or make dizzy (e.g., antidepressants, anti-seizure drugs)
* muscle disease (e.g., myasthenia gravis, myopathy, myositis)
* active hernia
* pregnancy
* muscle atrophy (e.g., Duchenne muscular dystrophy (DMD), Becker muscular dystrophy (BMD), ALS)
* neuro degenerative disease
* limited mobility
* those who consume proteins supplements.
* Individuals who have implanted pacemakers or defibrillators
* People who suffer from: Marfan syndrome, migraine, hyperparathyroidism, metastatic bone disease, multiple myeloma
* chronic steroid use
* individuals with restrictions to movement and exercise

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Lean Body Mass | 0-6 months
  Muscle measurements and fat composition will be assessed by Tanita at baseline (month 0) and month 6. Muscle mass, expressed as percentage change from baseline to month 6, will be compared within and between groups at 6 mos.
Body Circumference | 0-6 months
  Total body circumference will be measured by Army Body Fat Calculator at baseline (month 0) and month 6. Body circumference, expressed as percentage change from baseline to month 6, will be compared within and between groups at 6 mos.
Functional test 1 to assess musculoskeletal strength | 0-6 months
  Functional-Timed Up and Go Test will assess musculoskeletal strength at baseline (month 0) and month 6. Timed up-and-go times, expressed as change from baseline to month 6, will be compared within and between groups at 6 mos.
Functional test 2 to assess musculoskeletal strength | 0-6 months
  Functional-Sit-to-Stand Test will assess musculoskeletal strength at baseline (month 0) and month 6. Functional Sit-to-stand times, expressed as change from baseline to month 6, will be compared within and between groups at 6 mos.
Bone marker activity-bone resorption | 0-6 months
  Urinary CTx levels will be assessed at baseline (month 0) and month 6. The Effect of muscle strengthening on changes in Human Type 1 Collagen C-telopeptide (CTx) levels from baseline to month 6, will be compared within and between groups at 6 mos.
Bone marker activity-bone formation | 0-6 months
  Urinary P1NP levels will be assessed at baseline (month 0) and month 6. The Effect of muscle strengthening on changes in Human Procollagen Type 1 Intact N-terminal Propeptide (Total P1NP) levels from baseline will be compared within and between groups at 6 mos.
Ratio of bone resorption to bone formation | 0-6 months
  Urinary CTx:P1NP levels will be assessed at baseline (month 0) and month 6. The effect of muscle strengthening on changes in the ratio of CTx to P1NP will be assessed at baseline and then compared within and between groups at month 6.
Hormone levels-Testosterone | 0-6 months
  Urinary testosterone levels will be assessed at baseline (month 0) and month 6. The effect of muscle strengthening on changes in testosterone levels will be assessed at baseline and then compared within and between groups at month 6.
Hormone levels-Cortisol | 0-6 months
  Urinary cortisol levels will be assessed at baseline (month 0) and month 6. The effect of muscle strengthening on changes in cortisol levels will be assessed at baseline and then compared within and between groups at month 6.
Inflammatory Marker | 0-6 months
  Urinary C-reactive protein levels will be assessed at baseline (month 0) and then at month 6. The effect of muscle strengthening on changes in CRP will be assessed at baseline and then compared within and between groups at month 6.
Rest-activity rhythms | 0-6 months
  Rest activity rhythms will be assessed at baseline (month 0) and month 6. The effect of muscle strengthening on changes in rest-activity rhythms will be assessed at baseline and then compared within and between groups at month 6.
Melatonin | 0-6 months
  Salivary Melatonin levels will be assessed at baseline (month 0) and month 6. The effect of muscle strengthening on changes in melatonin rhythms will be assessed at baseline and then compared within and between groups at month 6.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Witt-Enderby, Ph.D., Principal Investigator — Duquesne University
Locations (1):
- Duquesne University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No